CLINICAL TRIAL: NCT06847932
Title: Leveraging AI-ECG Technology for Early Notification and Tracking of AF Development: a Randomized Control Trial
Brief Title: Leveraging AI-ECG Technology for Early Notification and Tracking of AF Development
Acronym: LATENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A202205179
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Premature Atrial Complexes; Atrial Arrhythmias; Artificial Intelligence (AI); Electrocardiogram
MeSH Terms: conditions — Atrial Fibrillation; Atrial Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF-predict AI-ECG alert system (Experimental): All the patients' ECGs will receive AF-predict AI-ECG analysis. According to the AI-ECG analysis results, those with at least one high-risk ECG within one year will be called back and asked to undergo a continuous cardiac rhythm monitor for up to 7 days. Otherwise, the physicians can review the AI-ECG analysis results for all the patients in the intervention group.
  Interventions: Other: AF-predict AI-ECG alert system guided management
- Standard of care (No Intervention): Patients will receive the standard care, and their ECGs will not be analyzed by AI-ECG before the end of the study.

INTERVENTIONS:
Other: AF-predict AI-ECG alert system guided management — AF-predict AI-ECG alert system
  Arms: AF-predict AI-ECG alert system

SUMMARY:
Our study aimed to use an AF-predict AI-ECG alert system to help physicians identify patients who need to wear a continuous cardiac rhythm monitor for new diagnoses of atrial fibrillation (AF), atrial flutter (AFL), or atrial arrhythmia with high AF risk, including premature atrial complexes (PAC) ≥ 500/24hr, burst PACs > 20 beats, non-sustained AF/AFL.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the inpatient department or the outpatient department
* Patients need to have at least one electrocardiogram within one year

Exclusion Criteria:

* Diagnosis of atrial fibrillation/atrial flutter
* History of atrial fibrillation/atrial flutter catheter ablation
* Patients with cardiac implantable electronic devices
* Any documented electrocardiogram showed atrial fibrillation/atrial flutter and pacing rhythm
* History of received rhythm control medications for atrial arrhythmia, including Class I and Class III antiarrhythmic drugs
* Any reasons indicate for anti-coagulant agents, including vitamin K antagonist and non-vitamin K antagonist oral anticoagulant

Ages: 40 Days to 85 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14726 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Latent atrial fibrillation | Within 90 days after enrollment.
  The primary outcome, latent atrial fibrillation, is a composite of new diagnoses of AF/AFL, atrial arrhythmia with high AF risk, including PACs ≥ 500/24hr, burst PACs > 20 beats, and non-sustained AF/AFL, within 90 days after enrollment. The results will be demonstrated as the rate of diagnoses of latent atrial fibrillation.

SECONDARY OUTCOMES:
Antiarrhythmic treatment | Within 180 days after enrollment.
  Antiarrhythmic treatment may include newly prescribed beta-blockers or non-dihydropyridine calcium channel blockers, class Ia, Ic, and III antiarrhythmic drugs, and catheter ablation. Physicians can determine whether a patient requires antiarrhythmic treatment through clinical practice. The outcome is the rate of initiation of antiarrhythmic treatment.
90-days New diagnoses of atrial fibrillation/atrial flutter | Within 90 days after enrollment.
  New diagnoses of atrial fibrillation or atrial flutter are defined as those documented by a 12-lead electrocardiogram or by continuous cardiac rhythm monitoring for ≥ 30 seconds. The result will be presented as the rate of new diagnoses of atrial fibrillation or atrial flutter.
Atrial arrhythmia with high AF risk | Within 90 days after enrollment.
  Atrial arrhythmia with high AF risk is defined by the following criteria: premature atrial complexes more than 500 beats in 24 hours as recorded by a continuous cardiac rhythm monitor; burst premature atrial complexes exceeding 20 beats as documented in a continuous cardiac rhythm monitor or a 12-lead electrocardiogram, or documented non-sustained AF/AFL in either a continuous cardiac rhythm monitor or a 12-lead electrocardiogram. The result will be presented as the rate of diagnoses of atrial arrhythmia with high AF risk.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lin, PhD, Principal Investigator — National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No